CLINICAL TRIAL: NCT06349707
Title: Relevance of the Multiplex PCR Approach for Severe Respiratory Infections of Patients Hospitalized - Including an Intensive Care Unit, During the COVID-19 Pandemic
Brief Title: Multiplex PCR for Severe Respiratory Infections During the COVID-19 Pandemic
Acronym: VirCoV+
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2023PI112
Record Dates: First submitted 2024-04-04; First posted 2024-04-05 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-04

CONDITIONS: Viral Pneumonia
Keywords: respiratory virus
MeSH Terms: conditions — Pneumonia, Viral

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18 ICU-patients group: 18 ICU (Intensive Care Unit)-patients group, from the whole population of patients (1,614) who were hospitalized for respiratory infections from early 2021 to mid-2022 in Nancy University hospital, France.
  Interventions: Other: other: Observational

INTERVENTIONS:
Other: other: Observational — For 18 ICU patients, retrospective collection of routine bioclinical database (ICCA db)

SUMMARY:
The hypothesis was that a retrospective investigation of the molecular virological tests in a University hospital could be informative, with the aim to identify non-COVID-19 respiratory viruses during the circulation of SARS-CoV-2, according to systematic population data for public health knowledge.

DETAILED DESCRIPTION:
The hypothesis was that a retrospective investigation of the molecular virological tests in a University hospital could be informative, with the aim to identify non-COVID-19 respiratory viruses during the circulation of SARS-CoV-2, according to systematic population data for public health knowledge:

* the main goal was to perform a retrospective investigation of the molecular virological tests in a University hospital, in order to identify non-COVID-19 respiratory viruses from the beginning of 2021 to mid-2022 during the circulation of SARS-CoV-2, for public health knowledge;
* the secondary aim was to retrospectively analyze, for a small subgroup of patients from an intensive care unit, the files of patients with positive molecular virological tests for non-COVID-19 respiratory viruses from the beginning of 2021 to mid-2022, reporting the following standard-of-care data: (i) the identification of the viruses, (ii) bioclinical features, (iii) medical impact of virological results in real life.

ELIGIBILITY:
Inclusion Criteria:

* For adult patients, or minors 'via' parents, able to give consent - 18 intensive care patients

Exclusion Criteria:

* Non-inclusion in case of refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 18 Intensive Care Unit (ICU)-patients, from the whole population of patients who were hospitalized for respiratory infections from early 2021 to mid-2022 in Nancy University hospital, France:
  * from the results of the multiplex FilmArrays PCR tests carried out during the 18 months of the study;
  * for the ICU files, 18 patients positive for virus by the FilmArray Pneumonia test: ICU patients (or representatives) informed of the data collection that can be used for research (ICCA db)
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of positive viral PCR assays (not COVID-19) from hospitalizations for respiratory infections. | 18 months, retrospectively
  Number of patients with positive virological molecular tests (multiplex respiratory panels) from the beginning of 2021 to mid-2022, with the nature of the viruses detected and the chronology of occurrence of positive tests.

SECONDARY OUTCOMES:
Real-life features of patients in Intensive care (from the whole population - Outcome 1) with positive viral PCR during infectious pneumonia. | 18 months, retrospectively
  For the group of patients in Intensive Care:
  * (i) number of positive molecular virological tests detecting respiratory viruses by FilmArray Pneumonia test
  * (ii) associated bioclinical data
  * (iii) medical impact of virological results in real life - progression of the infection and duration of thehospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Schvoerer, Vandœuvre-lès-Nancy, France